CLINICAL TRIAL: NCT01916798
Title: Intravenous Intralipid Therapy Among Women Aged 35-40 Years With Positive Peripheral Blood Natural Killer Cells Undergoing in Vitro Fertilization-Embryo Transfer: A Randomized Controlled Trial.
Brief Title: Intralipid Therapy for Women 35-40 Years With Positive Natural Killer Cells Undergoing Intracytoplasmic Sperm Injection (ICSI)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not able to recruit the number required and due to financial difficulty to pay for intralipids
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Elkattan, Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 300
Record Dates: First submitted 2013-08-03; First posted 2013-08-06 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Infertility
Keywords: Infertility; intralipid; invitro fertilization; repeated implantation failure; repeated miscarriage
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intralipid infusion (Active Comparator): 100 Subfertile women aged 35-40 years with repeated implantation failure or recurrent miscarriage with positive natural killer cells undergoing ICSI cycle.
  Interventions: Drug: Intralipid infusion
- Control group (No Intervention): 100 Subfertile women aged 35-40 years with repeated implantation failure or recurrent miscarriage with positive natural killer cells undergoing ICSI cycle.

INTERVENTIONS:
Drug: Intralipid infusion — IV infusion of 250 ml of intralipid 20% solution at the day of Ovum pick up & another dose at the day of embryo Transfer.
  Arms: Intralipid infusion

SUMMARY:
Intralipid can suppress natural killer cells that are known to be involve in repeated implantation failure and recurrent miscarriages.Intralipid is made of purified soybean oil, egg phospholipids, glycerol and water. It provides essential fatty acids, linoleic acid, omega- 3 and 6 fatty acids and alpha-linolenic acid. The effects of Intralipid in suppressing natural killer cell activity (NKa) were found to be comparable to intravenous immunoglobulin (IVIG) by laboratory experiments.We will study the effect of intralipid infusion on the pregnancy outcome of women aged 35-40 years with history of repeated implantation failure of miscarriage and who have positive peripheral blood natural killer cells

ELIGIBILITY:
Inclusion Criteria:

Subfertile women aged 35-40 years with repeated implantation failure or recurrent miscarriage with positive natural killer cells undergoing Intracytoplasmic sperm injection (ICSI ) cycle.

Exclusion Criteria:

* women above 40years or less than 35 years
* Disturbances of normal fat metabolism such as pathologic hyperlipidemia,Lipoid nephrosis or acute pancreatitis with hyperlipidemia.
* Allergic to eggs, soybean oil, or safflower oil.
* Severe liver disease, kidney disease, lung disease, anemia, blood coagulation disorder.
* Uterine fibroid, endometrial polyp, endometriosis and hydrosalpinx.
* Antiphospholipid syndrome (lupus anticoagulant and/or anticardiolipin antibodies (Immunoglobulin G or M)[IgG or IgM]); other recognised thrombophilic conditions (testing according to usual clinic practice).
* Intrauterine abnormalities (as assessed by ultrasound, hysterosonography, hysterosalpingogram, or hysteroscopy).
* Fibroids distorting uterine cavity.
* Abnormal parental karyotype.

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 10 months
  Intrauterine gestational sac with fatal pole and positive pulsation

SECONDARY OUTCOMES:
Chemical pregnancy | 10 months
  positive pregnancy test (serum BHCG) measured 16 days following embryo transfer
implantation rate | 10 months
  the number of gestational sacs divided by the number of embryos transferred
ongoing pregnancy rate | 10 months
  clinical pregnancy continue after 12 weeks gestational age
Miscarriage rate | 12 months
Ectopic rate | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Coulam CB, Acacio B. Does immunotherapy for treatment of reproductive failure enhance live births? Am J Reprod Immunol. 2012 Apr;67(4):296-304. doi: 10.1111/j.1600-0897.2012.01111.x. Epub 2012 Feb 16. PMID 22340745
- [Background] Shreeve N, Sadek K. Intralipid therapy for recurrent implantation failure: new hope or false dawn? J Reprod Immunol. 2012 Jan;93(1):38-40. doi: 10.1016/j.jri.2011.11.003. Epub 2011 Dec 21. PMID 22196107